CLINICAL TRIAL: NCT02074280
Title: Rifaximin Predicts the Complications of Decompensated Cirrhosis: a Randomized Controlled Trial
Brief Title: Rifaximin Predicts the Complications of Decompensated Cirrhosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Wei-Fen Xie, Director, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LPDLCC-1
Record Dates: First submitted 2014-02-15; First posted 2014-02-28 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Cirrhosis
Keywords: rifaximin; endotoxemia; cirrhosis; advanced cirrhosis
MeSH Terms: conditions — Fibrosis; Endotoxemia | interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- high dose of rifaximin (Experimental): rifaximin 600 mg, bid, orally, 2 weeks and conventional treatment
  Interventions: Drug: rifaximin
- low dose of rifaximin (Experimental): rifaximin 400 mg bid,orally, 2 weeks
  Interventions: Drug: rifaximin
- control (No Intervention): conventional treatment

INTERVENTIONS:
Drug: rifaximin — Rifaximin is an antibiotic that is virtually non-absorbed after oral administration and exhibits broad spectrum antimicrobial activity against both aerobic and anaerobic gram-positive and gram-negative microorganisms within the gastrointestinal tract.
  Arms: high dose of rifaximin; low dose of rifaximin

SUMMARY:
Cirrhotic patients are predisposed to intestinal dysmotility, bacterial overgrowth, and increased intestinal permeability all leading to an increase in bacterial translocation and increased endotoxemia. Rifaximin is an antibiotic that is virtually non-absorbed after oral administration and exhibits broad spectrum antimicrobial activity against both aerobic and anaerobic gram-positive and gram-negative microorganisms within the gastrointestinal tract. It has been suggested that oral prophylactic antibiotics or bowel decontamination might improve long-term outcomes in patients with cirrhosis. The aim of this study was to explore the suitable dose of rifaximin to alleviate endotoxemia and prevent the complications of advanced cirrhosis.

DETAILED DESCRIPTION:
Cirrhotic patients are predisposed to intestinal dysmotility, bacterial overgrowth, and increased intestinal permeability all leading to an increase in bacterial translocation and increased endotoxemia. Cirrhotics with bacterial translocation and endotoxemia manifest hemodynamic derangement with lower systemic vascular resistance, higher cardiac output, and lower mean arterial pressure. Moreover, endotoxins may increase portal pressure by increasing vascular resistance which may be promoted through the cytokine-stimulated intrahepatic release of endothelin and cyclo-oxygenase products.

Indeed, bacterial infections are common in cirrhotic patients and have approximately 30% mortality at one month and a further 30% mortality at 12 months as documented in a systematic review comprising almost 12 000 patients. It follows that altering gut flora to decrease endotoxin levels may lead to improved prognosis in cirrhosis. Rifaximin is an antibiotic that is virtually non-absorbed after oral administration and exhibits broad spectrum antimicrobial activity against both aerobic and anaerobic gram-positive and gram-negative microorganisms within the gastrointestinal tract. It has been suggested that oral prophylactic antibiotics or bowel decontamination might improve long-term outcomes in patients with cirrhosis, not only by reducing the risk of infections but also by reducing hepatic vein pressure gradient (HVPG).

The aim of this study was to explore the suitable dose of rifaximin to alleviate endotoxemia and prevent the complications of advanced cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Decompensated cirrhosis
* Child-Pugh B or C stage

Exclusion Criteria:

* severe complications of cirrhosis in the past one month.
* renal dysfunction.
* administration of antibiotics in the past two weeks.
* malignant tumors.
* HIV infection.
* severe heart and lung disease
* sensitivity to rifaximin
* Pregnancy and lactation woman
* Patients who have took part in other clinical trials in the past three months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Serum endotoxin level | 4 weeks
Hydrogen breath test | 4 weeks
Fecal flora | 4 weeks

SECONDARY OUTCOMES:
Liver biochemistry tests | 4 weeks
Numbers of complications of cirrhosis | 4 weeks
Serum levels of inflammatory factors | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Fen Xie, MD, Principal Investigator — Department of Gastroenterology, Changzheng Hospital, Second Military Medical University Shanghai
Locations (1):
- Shanghai changzheng Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Mullen KD, Sanyal AJ, Bass NM, Poordad FF, Sheikh MY, Frederick RT, Bortey E, Forbes WP. Rifaximin is safe and well tolerated for long-term maintenance of remission from overt hepatic encephalopathy. Clin Gastroenterol Hepatol. 2014 Aug;12(8):1390-7.e2. doi: 10.1016/j.cgh.2013.12.021. Epub 2013 Dec 21. PMID 24365449
- [Background] Xu D, Gao J, Gillilland M 3rd, Wu X, Song I, Kao JY, Owyang C. Rifaximin alters intestinal bacteria and prevents stress-induced gut inflammation and visceral hyperalgesia in rats. Gastroenterology. 2014 Feb;146(2):484-96.e4. doi: 10.1053/j.gastro.2013.10.026. Epub 2013 Oct 22. PMID 24161699
- [Background] Lutz P, Parcina M, Bekeredjian-Ding I, Hoerauf A, Strassburg CP, Spengler U. Spontaneous bacterial peritonitis by Pasteurella multocida under treatment with rifaximin. Infection. 2014 Feb;42(1):175-7. doi: 10.1007/s15010-013-0449-4. Epub 2013 Mar 25. PMID 23526308